CLINICAL TRIAL: NCT03375281
Title: Radiofrequency Ablation Using Octopus Electrodes for Small Hepatocellular Carcinoma With No-touch Technique: A Prospective Single Arm Study
Brief Title: Radiofrequency Ablation Using Octopus Electrodes for Small Hepatocellular Carcinoma With No-touch Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Starmed (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUH-2017-0870
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Hepatocellular Carcinoma; Radiofrequency Ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No touch group (Experimental): RFA for small HCC would be done by using no touch technique
  Interventions: Procedure: RFA

INTERVENTIONS:
Procedure: RFA — thermal ablation using radiofrequency for HCC

SUMMARY:
The aim of this study is to evaluate clinical outcome of RFA for small single nodular HCC using no touch technique with separable clustered electrode (Octopus) in a prospective multicenter manner Participating center: Seoul national university hospital, Asan medical center, Samsung medical center, Kunkuk university hospital, St. mary's Seoul hospital

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh class A liver function
* 1 - 2.5 cm sized Single nodular HCC
* without history of previous HCC treatment or with evidence of no recurrence at least 2 years after previous HCC treatment

Exclusion Criteria:

* more than 2 HCC
* tumor size larger than 2.5 cm
* Child-Pugh class B or C liver function
* invisible tumor even after real-time fusion US guidance
* accompanied by vascular invasion or distant metastasis
* presence of coagulopathy defined as platelet count < 50,000/mm3 and/or PT-INR > 50%

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
1 year local tumor progression | 1 year after procedure
  cumulative incidence of local tumor progression after RFA

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, M.D., Principal Investigator — Seoul National University Hospital
Locations (5):
- South Korea (5):
  - Asan medical Center, Seoul
  - Samsung medical center, Seoul
  - KonKuk university hospital, Seoul
  - Saint Mary Hospital, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee DH, Lee MW, Kim PN, Lee YJ, Park HS, Lee JM. Outcome of No-Touch Radiofrequency Ablation for Small Hepatocellular Carcinoma: A Multicenter Clinical Trial. Radiology. 2021 Oct;301(1):229-236. doi: 10.1148/radiol.2021210309. Epub 2021 Jul 27. PMID 34313474